CLINICAL TRIAL: NCT05195918
Title: Dose Ranging Study of Oral Epigallocatechin-3-gallate (EGCG) Given Daily for 12 Weeks to Patients With Idiopathic Pulmonary Fibrosis (IPF) Evaluating Safety, PK Interactions With Standard of Care Drugs, and Biomarkers of Drug Effect
Brief Title: Study of Oral Epigallocatechin-3-gallate (EGCG) in IPF Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hal Chapman (Other)
Collaborators: University of Michigan (Other); Cornell University (Other); Massachusetts General Hospital (Other); Temple University (Other); University of Washington (Other); University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Hal Chapman, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-35979
Record Dates: First submitted 2021-12-02; First posted 2022-01-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; epigallocatechin-3-gallate; EGCG
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — epigallocatechin gallate; nintedanib; pirfenidone

STUDY DESIGN:
Intervention Model Description: There will be two stages in this multi-center, double-blind, placebo-controlled, dose-ranging Phase I study. Participants will first be randomized to one of the four groups to receive 300 mg EGCG or placebo with one of the standard of care drugs (nintedanib or pirfenidone) for 12 weeks and 4 weeks follow-up. Once all 25 subjects at stage one have completed the study, a staged safety analysis will occur prior to opening stage two study with a higher group dose of 600 mg EGCG.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will be on one of the standard of care drugs (nintedanib or pirfenidone) and blindly given EGCG or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- EGCG 300 mg with Nintedanib (Active Comparator): Patients enrolled in this group will be given oral capsule EGCG 300 mg daily with doctor provided Nintedanib for 12 weeks.
  Interventions: Combination Product: EGCG 300 mg + Nintedanib
- EGCG 300 mg with Pirfenidone (Active Comparator): Patients enrolled in this group will be given oral capsule EGCG 300 mg daily with doctor provided Pirfenidone for 12 weeks.
  Interventions: Combination Product: EGCG 300 mg + Pirfenidone
- Placebo for EGCG 300 mg (Placebo Comparator): Patients enrolled in this group will be given oral capsule Placebo daily for 12 weeks with doctor provided Nintedanib or Pirfenidone. The number of placebo capsules will be equal to that of 300 mg EGCG.
  Interventions: Combination Product: Placebo 2 capsules + Nintedanib or Pirfenidone
- EGCG 600 mg with Nintedanib (Active Comparator): Patients enrolled in this group will be given oral capsule EGCG 600 mg daily with doctor provided Nintedanib for 12 weeks.
  Interventions: Combination Product: EGCG 600 mg + Nintedanib
- EGCG 600 mg with Pirfenidone (Active Comparator): Patients enrolled in this group will be given oral capsule EGCG 300 mg daily with doctor provided Pirfenidone for 12 weeks.
  Interventions: Combination Product: EGCG 600 mg + Pirfenidone
- Placebo for EGCG 600 mg (Placebo Comparator): Patients enrolled in this group will be given oral capsule Placebo daily for 12 weeks with doctor provided Nintedanib or Pirfenidone. The number of placebo capsules will be equal to that of 600 mg EGCG.
  Interventions: Combination Product: Placebo 4 capsules + Nintedanib or Pirfenidone

INTERVENTIONS:
Combination Product: EGCG 300 mg + Nintedanib — Dietary Supplement: EGCG Capsules with Teavigo EGCG (at least 94% purity). 300 mg EGCG (2 capsules) taken orally daily for 12 weeks.
  Drug: Nintedanib
  Other Names: epigallocatechin-3-gallate + Ofev
  Arms: EGCG 300 mg with Nintedanib
Combination Product: EGCG 300 mg + Pirfenidone — Dietary Supplement: EGCG Capsules with Teavigo EGCG (at least 94% purity). 300 mg EGCG (2 capsules) taken orally daily for 12 weeks.
  Drug: Pirfenidone
  Other Names: epigallocatechin-3-gallate + Esbriet
  Arms: EGCG 300 mg with Pirfenidone
Combination Product: Placebo 2 capsules + Nintedanib or Pirfenidone — Dietary Supplement: Placebo Placebo (2 capsules) taken orally daily for 12 weeks.
  Drug: Nintedanib
  Drug: Pirfenidone
  Other Names: Placebo + Ofev or Esbriet
  Arms: Placebo for EGCG 300 mg
Combination Product: EGCG 600 mg + Nintedanib — Dietary Supplement: EGCG Capsules with Teavigo EGCG (at least 94% purity). 600 mg EGCG (2 capsules) taken orally daily for 12 weeks.
  Drug: Nintedanib
  Other Names: epigallocatechin-3-gallate + Ofev
  Arms: EGCG 600 mg with Nintedanib
Combination Product: EGCG 600 mg + Pirfenidone — Dietary Supplement: EGCG Capsules with Teavigo EGCG (at least 94% purity). 600 mg EGCG (2 capsules) taken orally daily for 12 weeks.
  Drug: Pirfenidone
  Other Names: epigallocatechin-3-gallate + Esbriet
  Arms: EGCG 600 mg with Pirfenidone
Combination Product: Placebo 4 capsules + Nintedanib or Pirfenidone — Dietary Supplement: Placebo Placebo (4 capsules) taken orally daily for 12 weeks.
  Drug: Nintedanib
  Drug: Pirfenidone
  Other Names: Placebo + Ofev or Esbriet
  Arms: Placebo for EGCG 600 mg

SUMMARY:
The primary purpose of this multi-center, double-blind, placebo-controlled, dose-ranging Phase I study is to assess the safety of a purified from green tea, EGCG, in patients with idiopathic pulmonary fibrosis (IPF) as a potential novel treatment for pulmonary fibrosis.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, placebo-controlled, dose-ranging Phase I study of once daily EGCG administered for 12 weeks. The study will assess safety, pharmacokinetics, and biomarker measurements of drug effect in IPF patients already receiving background therapy for IPF with either nintedanib or pirfenidone. Two different doses of EGCG will be studied.

The rationale for this study is 1) extensive pre-clinical data in mice that EGCG is efficacious in attenuating pulmonary fibrosis by blocking collagen cross-linking and the pro-fibrotic pathway mediated by TGFβ1 signaling and 2) recently published data demonstrating that in humans EGCG is safe and capable of blocking lung tissue pro-fibrotic signaling when given two weeks prior to diagnostic surgical biopsy of pulmonary fibrosis patients, many of whom were subsequently diagnosed with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 40-85 years old.
4. Participant has IPF satisfying the 2022 ATS diagnostic criteria, confirmed by enrolling investigator at Visit 1.
5. Participant must have been on a stable dose of nintedanib twice daily or pirfenidone three times daily dose for at least 12 weeks prior to baseline (Visit 2).
6. Participant has a FVC ≥ 50% predicted using the global lung function initiative (GLI).
7. Participant has a DLCO corrected for hemoglobin ≥ 35% predicted using the GLI.
8. Women of child bearing potential (WCBP), defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if < 55 years or 12 months if > 55 years, must have a negative serum pregnancy test within 1 week prior to the first dose of study drug and must agree to use adequate methods of birth control throughout the study. Adequate methods of contraception include use of oral contraceptives or Depo-Provera, with an additional barrier method (diaphragm with spermicidal gel or condoms with spermicide), double-barrier methods (diaphragm with spermicidal gel and condoms with spermicide), partner vasectomy, and total abstinence.
9. Participant has a life expectancy of at least 9 months at Visit 1.
10. Ability to take oral medication and be willing to adhere to EGCG regimen.
11. Agreement to refrain from drinking green tea in excess of a cup a day or eating green tea extract for 4 weeks before baseline and during the trial.

Exclusion Criteria:

1. AST, ALT, or direct bilirubin above upper limit normal from any cause at the Screening Visit.
2. Any history of HCV or HBV infection, NASH/NAFLD, or cirrhosis.
3. Alcohol consumption greater than 7 drinks per week.
4. Participant has emphysema ≥ 50% or the extent of emphysema is greater than the extent of fibrosis as per interpretation of Site Investigator or radiologist.
5. Participant has received investigational therapy for IPF within 4 weeks before baseline (Visit 2).
6. Participant is receiving systemic corticosteroids equivalent to prednisone > 10 mg/day or equivalent within 2 weeks of baseline visit (Visit 2).
7. Participant has any concurrent condition other than IPF that, in the Investigator's opinion, is unstable and/or would impact the likelihood of survival for the study duration or the participant's ability to complete the study as designed, or may influence any of the safety or efficacy assessments included in the study.
8. Participant has baseline resting oxygen saturation of < 89% on room air or need for continuous oxygen use at baseline visit (Visit 2).
9. Consumption of GTE products in excess of a cup of green tea a day within one month of the baseline visit (Visit 2).
10. Participant is receiving digoxin at the time of screening (Visit 1) and for the duration of the study.
11. Active respiratory infection requiring treatment with antibiotics within 4 weeks of the baseline visit (Visit 2).
12. Likely to be listed for transplant during trial participation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Participants with treatment-emergent adverse event (TEAE) | Up to 12 weeks
  The number of participants with at least 1 treatment-emergent adverse event
The number of treatment-emergent adverse events (TEAE) | Up to 12 weeks
  The number of treatment-emergent adverse events
Participants with grade 3 or 4 treatment-emergent adverse events (TEAE) | Up to 12 weeks
  The number of participants with at least 1 grade 3 or 4 treatment-emergent adverse events
The number of grade 3 or 4 treatment-emergent adverse events (TEAE) | Up to 12 weeks
  The number of grade 3 or 4 treatment-emergent adverse events
Participants with serious adverse event (SAE) | Up to 12 weeks
  The number of participants with at least 1 serious adverse event
The number of serious adverse event (SAE) | Up to 12 weeks
  The number of serious adverse events
Participants with discontinued study treatment due to adverse events (AE) | Up to 12 weeks
  The number of participants who discontinued study treatment due to adverse events
Participants with discontinued study treatment due to serious adverse events (SAE) | Up to 12 weeks
  The number of participants who discontinued study treatment due to serious adverse events
Participants died due to adverse events (AE) on study treatment | Up to 12 weeks
  The number of participants who died due to adverse events on study treatment
Participants died due to adverse events (AE) within 4 weeks of discontinuation | Up to 12 weeks
  The number of participants who died due to adverse events within 4 weeks of discontinuation from study treatment
Participants with adverse event (AE) by causality | Up to 12 weeks
  The number of participants with at least 1 adverse event by causality (reasonable possibility/no reasonable possibility)
Adverse events (AE) by causality | Up to 12 weeks
  The number of adverse events by causality (reasonable possibility/no reasonable possibility)
Change in individual laboratory parameters | Up to 12 weeks
  Absolute and relative change in individual laboratory parameters from baseline at day 84
Change in forced vital capacity (FVC) | Up to 12 weeks
  Absolute and relative change in forced vital capacity from baseline at day 84
Change in forced vital capacity (FVC) % predicted | Up to 12 weeks
  Absolute and relative change in forced vital capacity % predicted from baseline at day 84
Change in diffusing capacity for carbon monoxide (DLCO) | Up to 12 weeks
  Absolute and relative change in diffusing capacity for carbon monoxide uncorrected for hemoglobin from baseline at day 84
Change in total score for the King's Brief Interstitial Lung Disease (K-BILD) Questionnaire | Up to 12 weeks
  Absolute change in total score for the King's Brief Interstitial Lung Disease (K-BILD) Questionnaire from baseline at day 84
Participants with an absolute change in K-BILD of 5 points or more in either direction | Up to 12 weeks
  The number of participants with an absolute change in K-BILD from baseline to day 84 of 5 points or more in either direction
Change in total score for the Leicester Cough Questionnaire (LCQ) | Up to 12 weeks
  Absolute change in total score for the Leicester Cough Questionnaire (LCQ) from baseline at day 84
Participants with an absolute change of at least 1.5 points for the LCQ | Up to 12 weeks
  The number of participants with an absolute change from baseline to day 84 of 1.5 points or more in either direction for the LCQ
Participants with a peak level change for nintedanib or pirfenidone over 50% from screening to baseline (day 1) | Day 1
  The number of participants with a change from screening to baseline (day 1) in peak levels for nintedanib or pirfenidone of 50% or more in either direction
Participants with a peak level change for nintedanib or pirfenidone over 50% from baseline to day 14 | Day 14
  The number of participants with a change from baseline to day 14 in peak levels for nintedanib or pirfenidone of 50% or more in either direction
Participants with a trough level change for nintedanib or pirfenidone over 50% from baseline to day 14 | Day 14
  The number of participants with a change from baseline to day 14 in trough levels for nintedanib or pirfenidone of 50% or more in either direction
Participants with peak (cmax) levels for EGCG < 250 nM at day 14 | Day 14
  The number of participants with peak (cmax) levels for EGCG < 250 nM at day 14

SECONDARY OUTCOMES:
Change of serum biomarker COMP at day 14 | Day 14
  Change in level of serum biomarker COMP from baseline at day 14
Change of serum biomarker COMP at day 84 | Day 84
  Change in level of serum biomarker COMP from baseline at day 84
Change of serum biomarker Periostin at day 14 | Day 14
  Change in level of serum biomarker Periostin from baseline at day 14
Change of serum biomarker Periostin at day 84 | Day 84
  Change in level of serum biomarker Periostin from baseline at day 84
Change of serum biomarker pro-MMP1 at day 14 | Day 14
  Change in level of serum biomarker pro-MMP1 from baseline at day 14
Change of serum biomarker pro-MMP1 at day 84 | Day 84
  Change in level of serum biomarker pro-MMP1 from baseline at day 84

CONTACTS AND LOCATIONS:
Overall Officials: Harold Chapman, MD, Principal Investigator — University of California, San Francisco; Fernando J Martinez, MD, Principal Investigator — Cornell University; Sydney Montesi, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - UCSF Parnassus, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medicine, New York, New York
  - Temple University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei Y, Kim TJ, Peng DH, Duan D, Gibbons DL, Yamauchi M, Jackson JR, Le Saux CJ, Calhoun C, Peters J, Derynck R, Backes BJ, Chapman HA. Fibroblast-specific inhibition of TGF-beta1 signaling attenuates lung and tumor fibrosis. J Clin Invest. 2017 Oct 2;127(10):3675-3688. doi: 10.1172/JCI94624. Epub 2017 Sep 5. PMID 28872461
- [Background] Raghu G, Brown KK, Collard HR, Cottin V, Gibson KF, Kaner RJ, Lederer DJ, Martinez FJ, Noble PW, Song JW, Wells AU, Whelan TP, Wuyts W, Moreau E, Patterson SD, Smith V, Bayly S, Chien JW, Gong Q, Zhang JJ, O'Riordan TG. Efficacy of simtuzumab versus placebo in patients with idiopathic pulmonary fibrosis: a randomised, double-blind, controlled, phase 2 trial. Lancet Respir Med. 2017 Jan;5(1):22-32. doi: 10.1016/S2213-2600(16)30421-0. Epub 2016 Dec 7. PMID 27939076
- [Background] Hu J, Webster D, Cao J, Shao A. The safety of green tea and green tea extract consumption in adults - Results of a systematic review. Regul Toxicol Pharmacol. 2018 Jun;95:412-433. doi: 10.1016/j.yrtph.2018.03.019. Epub 2018 Mar 24. PMID 29580974
- [Background] Isomura T, Suzuki S, Origasa H, Hosono A, Suzuki M, Sawada T, Terao S, Muto Y, Koga T. Liver-related safety assessment of green tea extracts in humans: a systematic review of randomized controlled trials. Eur J Clin Nutr. 2016 Nov;70(11):1221-1229. doi: 10.1038/ejcn.2016.78. Epub 2016 May 18. PMID 27188915
- [Background] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133
- [Background] Corte T, Bonella F, Crestani B, Demedts MG, Richeldi L, Coeck C, Pelling K, Quaresma M, Lasky JA. Safety, tolerability and appropriate use of nintedanib in idiopathic pulmonary fibrosis. Respir Res. 2015 Sep 24;16:116. doi: 10.1186/s12931-015-0276-5. PMID 26400368
- [Background] Li H, Chang HM, Shi Z, Leung PCK. ID3 mediates the TGF-beta1-induced suppression of matrix metalloproteinase-1 in human granulosa cells. FEBS J. 2019 Nov;286(21):4310-4327. doi: 10.1111/febs.14964. Epub 2019 Jun 28. PMID 31215762
- [Background] Sheppard D. Transforming growth factor beta: a central modulator of pulmonary and airway inflammation and fibrosis. Proc Am Thorac Soc. 2006 Jul;3(5):413-7. doi: 10.1513/pats.200601-008AW. PMID 16799084
- [Background] Principe DR, DeCant B, Mascarinas E, Wayne EA, Diaz AM, Akagi N, Hwang R, Pasche B, Dawson DW, Fang D, Bentrem DJ, Munshi HG, Jung B, Grippo PJ. TGFbeta Signaling in the Pancreatic Tumor Microenvironment Promotes Fibrosis and Immune Evasion to Facilitate Tumorigenesis. Cancer Res. 2016 May 1;76(9):2525-39. doi: 10.1158/0008-5472.CAN-15-1293. Epub 2016 Mar 15. PMID 26980767
- [Background] Ignotz RA, Massague J. Transforming growth factor-beta stimulates the expression of fibronectin and collagen and their incorporation into the extracellular matrix. J Biol Chem. 1986 Mar 25;261(9):4337-45. PMID 3456347
- [Background] Akhurst RJ, Hata A. Targeting the TGFbeta signalling pathway in disease. Nat Rev Drug Discov. 2012 Oct;11(10):790-811. doi: 10.1038/nrd3810. Epub 2012 Sep 24. PMID 23000686
- [Background] Lacouture ME, Morris JC, Lawrence DP, Tan AR, Olencki TE, Shapiro GI, Dezube BJ, Berzofsky JA, Hsu FJ, Guitart J. Cutaneous keratoacanthomas/squamous cell carcinomas associated with neutralization of transforming growth factor beta by the monoclonal antibody fresolimumab (GC1008). Cancer Immunol Immunother. 2015 Apr;64(4):437-46. doi: 10.1007/s00262-015-1653-0. Epub 2015 Jan 13. PMID 25579378
- [Background] Hu GX, Yao ST, Zeng LH, Peng YZ, Zheng J. Effects of hydroxycamptothecin on the expression of matrix metalloproteinase-1 (MMP-1), tissue inhibitor of MMP-1, and type I collagen in rats with pulmonary fibrosis. Genet Mol Res. 2015 May 4;14(2):4625-32. doi: 10.4238/2015.May.4.21. PMID 25966236
- [Background] Lee MJ, Maliakal P, Chen L, Meng X, Bondoc FY, Prabhu S, Lambert G, Mohr S, Yang CS. Pharmacokinetics of tea catechins after ingestion of green tea and (-)-epigallocatechin-3-gallate by humans: formation of different metabolites and individual variability. Cancer Epidemiol Biomarkers Prev. 2002 Oct;11(10 Pt 1):1025-32. PMID 12376503
- [Background] Li M, Krishnaveni MS, Li C, Zhou B, Xing Y, Banfalvi A, Li A, Lombardi V, Akbari O, Borok Z, Minoo P. Epithelium-specific deletion of TGF-beta receptor type II protects mice from bleomycin-induced pulmonary fibrosis. J Clin Invest. 2011 Jan;121(1):277-87. doi: 10.1172/JCI42090. Epub 2010 Dec 6. PMID 21135509
- [Background] Mereles D, Hunstein W. Epigallocatechin-3-gallate (EGCG) for clinical trials: more pitfalls than promises? Int J Mol Sci. 2011;12(9):5592-603. doi: 10.3390/ijms12095592. Epub 2011 Aug 31. PMID 22016611
- [Background] Mertens-Talcott SU, Jilma-Stohlawetz P, Rios J, Hingorani L, Derendorf H. Absorption, metabolism, and antioxidant effects of pomegranate (Punica granatum l.) polyphenols after ingestion of a standardized extract in healthy human volunteers. J Agric Food Chem. 2006 Nov 15;54(23):8956-61. doi: 10.1021/jf061674h. PMID 17090147
- [Background] Nagle DG, Ferreira D, Zhou YD. Epigallocatechin-3-gallate (EGCG): chemical and biomedical perspectives. Phytochemistry. 2006 Sep;67(17):1849-55. doi: 10.1016/j.phytochem.2006.06.020. Epub 2006 Jul 31. PMID 16876833
- [Background] Stoner GD, Sardo C, Apseloff G, Mullet D, Wargo W, Pound V, Singh A, Sanders J, Aziz R, Casto B, Sun X. Pharmacokinetics of anthocyanins and ellagic acid in healthy volunteers fed freeze-dried black raspberries daily for 7 days. J Clin Pharmacol. 2005 Oct;45(10):1153-64. doi: 10.1177/0091270005279636. PMID 16172180
- [Background] Chen Y, Guo H, Terajima M, Banerjee P, Liu X, Yu J, Momin AA, Katayama H, Hanash SM, Burns AR, Fields GB, Yamauchi M, Kurie JM. Lysyl Hydroxylase 2 Is Secreted by Tumor Cells and Can Modify Collagen in the Extracellular Space. J Biol Chem. 2016 Dec 9;291(50):25799-25808. doi: 10.1074/jbc.M116.759803. Epub 2016 Nov 1. PMID 27803159
- [Background] Zhang HM, Zhao L, Li H, Xu H, Chen WW, Tao L. Research progress on the anticarcinogenic actions and mechanisms of ellagic acid. Cancer Biol Med. 2014 Jun;11(2):92-100. doi: 10.7497/j.issn.2095-3941.2014.02.004. PMID 25009751
- [Background] Dostal AM, Samavat H, Bedell S, Torkelson C, Wang R, Swenson K, Le C, Wu AH, Ursin G, Yuan JM, Kurzer MS. The safety of green tea extract supplementation in postmenopausal women at risk for breast cancer: results of the Minnesota Green Tea Trial. Food Chem Toxicol. 2015 Sep;83:26-35. doi: 10.1016/j.fct.2015.05.019. Epub 2015 Jun 5. PMID 26051348
- [Background] Oketch-Rabah HA, Roe AL, Rider CV, Bonkovsky HL, Giancaspro GI, Navarro V, Paine MF, Betz JM, Marles RJ, Casper S, Gurley B, Jordan SA, He K, Kapoor MP, Rao TP, Sherker AH, Fontana RJ, Rossi S, Vuppalanchi R, Seeff LB, Stolz A, Ahmad J, Koh C, Serrano J, Low Dog T, Ko R. United States Pharmacopeia (USP) comprehensive review of the hepatotoxicity of green tea extracts. Toxicol Rep. 2020 Feb 15;7:386-402. doi: 10.1016/j.toxrep.2020.02.008. eCollection 2020. PMID 32140423
- [Background] Yu Z, Samavat H, Dostal AM, Wang R, Torkelson CJ, Yang CS, Butler LM, Kensler TW, Wu AH, Kurzer MS, Yuan JM. Effect of Green Tea Supplements on Liver Enzyme Elevation: Results from a Randomized Intervention Study in the United States. Cancer Prev Res (Phila). 2017 Oct;10(10):571-579. doi: 10.1158/1940-6207.CAPR-17-0160. Epub 2017 Aug 1. PMID 28765194
- [Background] Maher TM, Stowasser S, Nishioka Y, White ES, Cottin V, Noth I, Selman M, Rohr KB, Michael A, Ittrich C, Diefenbach C, Jenkins RG; INMARK trial investigators. Biomarkers of extracellular matrix turnover in patients with idiopathic pulmonary fibrosis given nintedanib (INMARK study): a randomised, placebo-controlled study. Lancet Respir Med. 2019 Sep;7(9):771-779. doi: 10.1016/S2213-2600(19)30255-3. Epub 2019 Jul 17. PMID 31326319
- [Background] Neighbors M, Cabanski CR, Ramalingam TR, Sheng XR, Tew GW, Gu C, Jia G, Peng K, Ray JM, Ley B, Wolters PJ, Collard HR, Arron JR. Prognostic and predictive biomarkers for patients with idiopathic pulmonary fibrosis treated with pirfenidone: post-hoc assessment of the CAPACITY and ASCEND trials. Lancet Respir Med. 2018 Aug;6(8):615-626. doi: 10.1016/S2213-2600(18)30185-1. Epub 2018 Jun 29. PMID 30072107
- [Result] Chapman HA, Wei Y, Montas G, Leong D, Golden JA, Trinh BN, Wolters PJ, Le Saux CJ, Jones KD, Hills NK, Foster E, Oldham JM, Linderholm AL, Kotak P, Decaris M, Turner S, Song JW. Reversal of TGFbeta1-Driven Profibrotic State in Patients with Pulmonary Fibrosis. N Engl J Med. 2020 Mar 12;382(11):1068-1070. doi: 10.1056/NEJMc1915189. No abstract available. PMID 32160670
- [Result] Wei Y, Dong W, Jackson J, Ho TC, Le Saux CJ, Brumwell A, Li X, Klesney-Tait J, Cohen ML, Wolters PJ, Chapman HA. Blocking LOXL2 and TGFbeta1 signalling induces collagen I turnover in precision-cut lung slices derived from patients with idiopathic pulmonary fibrosis. Thorax. 2021 Jul;76(7):729-732. doi: 10.1136/thoraxjnl-2020-215745. Epub 2021 Jan 20. PMID 33472968